CLINICAL TRIAL: NCT07108751
Title: Association Between Gastroesophageal Reflux Disease (GERD) Severity and Dental Caries: A Cross-Sectional Study
Brief Title: Association Between Gastroesophageal Reflux Disease (GERD) Severity and Dental Caries
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El-Raouf Tawfik, Professor of Internal Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR1280/7/25
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Gastroesophageal Reflux Disease; Severity; Dental Caries
MeSH Terms: conditions — Gastroesophageal Reflux; Dental Caries | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Gastroesophageal reflux disease (GERD) patients.
  Interventions: Device: Endoscopy
- Control group: Matched control group.
  Interventions: Device: Endoscopy

INTERVENTIONS:
Device: Endoscopy — Endoscopy will be performed to all patient

SUMMARY:
This study aimed to assess the relationship between gastroesophageal reflux disease (GERD) severity (based on upper gastrointestinal endoscopy) and dental caries severity.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a chronic condition characterized by reflux of stomach acid into the esophagus, with a prevalence reaching 20-30% in many populations. Beyond its gastrointestinal manifestations, GERD may have extraesophageal effects, including oral health disturbances such as dental erosion and caries. Exposure of the oral cavity to gastric acid, especially in patients with severe or nocturnal reflux, may contribute to enamel demineralization, increased tooth decay, and lower salivary pH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Both sexes.
* Diagnosed with Gastroesophageal Reflux Disease (GERD) by endoscopy.
* Consent to participate.

Exclusion Criteria:

* Xerostomia-related disorders.
* Recent antibiotics (last 4 weeks).
* Head/neck radiation history.
* Cognitive impairment affecting consent.
* Pregnant or lactating women.
* HbA1c above 6.4%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cross-sectional analytical study was conducted at the Gastrointestinal Endoscopy Unit of the Internal Medicine Department at Tanta University Hospital in Egypt, and the Outpatient Dental Clinic affiliated with Zarqa University Dental Clinics in Jordan between January and June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Decayed, Missing, and Filled Teeth (DMFT) Index | 3 months post-procedure
  The Decayed, Missing, and Filled Teeth (DMFT) Index was calculated as the sum of decayed, missing, and filled teeth, with scores ranging from 0 to 28 or 32, depending on the total number of teeth present.

SECONDARY OUTCOMES:
Basic Erosive Wear Examination Index | 3 months post-procedure
  The Basic Erosive Wear Examination Index was used to evaluate tooth surface erosion, with each of the six oral sextants scored based on the most severely affected tooth surface. Erosive wear was graded from 0 (no erosive wear) to 3 (hard tissue loss of 50 percent or greater of the surface area), with cumulative scores categorized into risk bands ranging from no risk (0-2) to high risk (≥14).
Plaque Index | 3 months post-procedure
  The Plaque Index was assessed by examining four surfaces per tooth (buccal, lingual, mesial, and distal) and scoring plaque thickness from 0 (no plaque) to 3 (heavy plaque accumulation), with final scores calculated as the total plaque scores divided by the number of surfaces examined.
Salivary analysis | 3 months post-procedure
  Saliva was accumulated in the mouth without stimulation and expectorated into sterile tubes every 60 seconds for five minutes. Salivary pH was measured immediately using a calibrated digital pH meter with measurements taken for 1-2 seconds in 1-2 mL samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.